CLINICAL TRIAL: NCT01724528
Title: Febuxostat for Tumor Lysis Syndrome Prevention in Hematologic Malignancies: a Randomized, Double Blind, Phase III Study Versus Allopurinol
Brief Title: Febuxostat for Tumor Lysis Syndrome Prevention in Hematologic Malignancies
Acronym: FLORENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLO-01; 2012-000776-42 (EudraCT Number)
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Tumor Lysis Syndrome
Keywords: Febuxostat, Tumor lysis syndrome, leukemia, lymphoma
MeSH Terms: conditions — Tumor Lysis Syndrome; Leukemia; Lymphoma | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Febuxostat (Experimental): Febuxostat for 7-9 days
  Interventions: Drug: Febuxostat
- Allopurinol (Active Comparator): Allopurinol for 7-9 days
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat — Standard dose PO (per os) from Day 1 to Day 7 (can be continued up to DAY 9 at investigator's discretion)
  Other Names: Adenuric
  Arms: Febuxostat
Drug: Allopurinol — Standard dose, low dose or high dose (as per investigator's judgement at the time of randomization) from DAY 1 to DAY 7 (can be continued up to DAY 9 at investigator's discretion)
  Other Names: Zyloric
  Arms: Allopurinol

SUMMARY:
The purpose of this study is to determine whether febuxostat is superior to allopurinol in the prevention of tumor lysis syndrome (TLS) in patients with hematological malignancies at intermediate or high risk of TLS (according to Cairo-Bishop classification) who undergo chemotherapy

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, active-controlled, parallel-group study to be conducted in approximately 80 sites.

Approximately 340 male or female patients aged 18 or older suffering from hematologic malignancies (de novo patients or relapsing patients) at intermediate to high risk of TLS and scheduled for receiving the first cycle of cytotoxic chemotherapy, regardless of the line of treatment, will be randomized in this study. Eligible patients (as per screening visit) will be randomly allocated in a 1:1 ratio to Febuxostat or Allopurinol. The double-blind treatment period starts two days prior to the planned beginning of chemotherapy and continues for 7 to 9 consecutive days, according to Investigator judgment and on the basis of the actual duration of chemotherapy regimen administered to the patient. Along the study treatment, uric acid levels, creatinine levels, Laboratory TLS/Clinical TLS and Adverse Events represent the major clinical findings to be monitored on a daily basis. Overall the study encompasses 10 to 11 planned visits at site, including screening, randomisation, on treatment and final follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first cytotoxic chemotherapy cycle, regardless of the line of treatment, because of hematologic malignancies at intermediate or high risk of TLS (according to the TLS risk stratification, Cairo M et al, British Journal of Haematology, 2010)candidate to Allopurinol treatment or have no access to Rasburicase
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3
* Life expectancy > 1 month

Exclusion Criteria:

* Patients known to be hypersensitive to Febuxostat or Allopurinol or to any of the components of the formulations
* Patients with sUA levels ≥ 10 mg/dL at randomization
* Patients receiving Febuxostat, Allopurinol or any other urate lowering therapy (e.g. Rasburicase, probenecid) within 30 days prior to randomization
* Patients with severe renal and/or hepatic insufficiency
* Patients with diagnosis of LTLS or CTLS at randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spina, MD, Principal Investigator — Centro Riferimento Oncologico (CRO) National Cancer Institute-Aviano-Italy; Angela Capriati, MD, PhD, Study Director — Menarini Ricerche S.p.A. - Florence-Italy

REFERENCES:
- [Derived] Spina M, Nagy Z, Ribera JM, Federico M, Aurer I, Jordan K, Borsaru G, Pristupa AS, Bosi A, Grosicki S, Glushko NL, Ristic D, Jakucs J, Montesinos P, Mayer J, Rego EM, Baldini S, Scartoni S, Capriati A, Maggi CA, Simonelli C; FLORENCE Study Group. FLORENCE: a randomized, double-blind, phase III pivotal study of febuxostat versus allopurinol for the prevention of tumor lysis syndrome (TLS) in patients with hematologic malignancies at intermediate to high TLS risk. Ann Oncol. 2015 Oct;26(10):2155-61. doi: 10.1093/annonc/mdv317. Epub 2015 Jul 27. PMID 26216382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in (screening) 01 Oct 2012, last patient out 11 Oct 2013. At 79 sites across 11 European countries (Croatia, Czech Republic, Germany, Hungary, Italy, Poland, Romania, Russia, Serbia, Spain and Ukraine) and Brazil
Pre-assignment Details: Subjects complying with inclusion/exclusion criteria were to be randomised to receive (blinded) standard, low or high dose of study treatment as per investigator's assessment (mainly based on renal function). Randomization was balanced by TLS risk and serum uric acid levels (≤ or > 7.5 mg/dL)
Period: Overall Study
Arm/Group | Febuxostat | Allopurinol
Started | 173 | 173
Completed | 169 | 170
Not Completed | 4 | 3
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Patient refused to attend last visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Allopurinol | Total
Number analyzed (Participants) | 173 | 173 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (14.26) | 58.3 (13.26) | 58.4 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 132
  Male | 108 | 106 | 214
serum uric acid (sUA) [Number; unit: participants]
  < or = 7.5 mg/dL | 151 | 152 | 303
  > 7.5 mg/dL | 22 | 21 | 43
TLS risk [Number; unit: participants]
  Intermediate | 143 | 141 | 284
  High | 30 | 32 | 62
Type of Hematologic Malignancy [Number; unit: participants]
  Acute leukemia | 34 | 25 | 59
  Chronic lymphocytic leukemia | 80 | 94 | 174
  Lymphoma | 59 | 54 | 113

OUTCOME MEASURES:

1. Primary Outcome: Serum Uric Acid (sUA) Level Control
Description: Area under the curve of sUA from baseline (Day 1) to the evaluation visit (Day 8)
Time Frame: 8 days
Population: Intention to treat (ITT), defined as all randomized patients. Sample size calculation: at least an absolute reduction of 100 mg x h/dL for the AUCsUA1-8 in favour of febuxostat; 340 patients were sufficient to achieve approximately 80% power. Imputation method: last observation carried forward (LOCF); missing baseline values were not replaced.
Measure: Mean (Standard Deviation); unit: mg x hour/dL
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 172 | 172
mg x hour/dL | 514.0 (225.71) | 708.0 (234.42)
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Treatment, TLS risk (intermediate/high) and sUA level at baseline (≤ 7.5 mg/dL and > 7.5 mg/dL) were inserted in the ANCOVA model as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares means difference = -196.794, 95% CI 2-sided [-238.600 to -154.988]

2. Primary Outcome: Preservation of Renal Function
Description: Change in serum creatinine level from baseline (Day 1) to the evaluation visit (Day 8)
Time Frame: 8 days
Population: ITT. Sample size calculation: no change in mean serum creatinine level from baseline to the end of treatment for febuxostat group while allopurinol has a increase of 13%; 340 patients were sufficient to achieve approximately 80% power. Imputation method: LOCF; missing baseline values were not replaced
Measure: Mean (Standard Deviation); unit: change %
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 173 | 171
change % | -0.83 (26.977) | -4.92 (16.695)
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0903, ANCOVA; Least squares means difference = 4.0970, 95% CI 2-sided [-0.6467 to 8.8406]

3. Secondary Outcome: Treatment Responder Rate
Description: Assessment of treatment responder rate, where treatment response is defined as the maintenance of sUA ≤ 7.5 mg/dL from Day 3 to Day 8
Time Frame: 6 days
Population: Intention to Treat (ITT; no imputation applied
Measure: Number; unit: % of patients who fail to respond
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 173 | 173
% of patients who fail to respond | 1.7 | 4.0
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.1993, Wilson's confidence interval; Risk Difference (RD) = 0.0231, 95% CI 2-sided [-0.0153 to 0.0654]

4. Secondary Outcome: Assessment of Laboratory Tumor Lysis Syndrome (LTLS)
Description: Assessment of LTLS, from Day 3 to Day 8. According to Cairo-Bishop definition LTLS is defined by the presence of 2 or more laboratory abnormalities including: a 25% increase or levels above normal for serum uric acid, potassium, and phosphate or a 25% decrease or levels below normal for calcium.
Time Frame: 6 days
Population: ITT; no imputation applied
Measure: Number; unit: % of patients with LTLS occurrence
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 173 | 173
% of patients with LTLS occurrence | 8.1 | 9.2
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 0.8488, Chi-squared; Relative risk = 0.875, 95% CI 2-sided [0.4408 to 1.7369]

5. Secondary Outcome: Assessment of Clinical Tumor Lysis Syndrome (CTLS)
Description: Assessment of CTLS, from Day 3 to Day 8. According to Cairo-Bishop definition, CTLS is defined by the presence of LTLS in addition to 1 or more of the following significant clinical complications: renal insufficiency, cardiac arrhythmias, sudden death and seizures. The grade of CTLS is defined by the maximal grade of the clinical manifestation
Time Frame: 6 days
Population: ITT; no imputation applied
Measure: Number; unit: % of patients with CTLS occurrence
Arm/Group | Febuxostat | Allopurinol
Number analyzed (Participants) | 173 | 173
% of patients with CTLS occurrence | 1.7 | 1.2
Statistical Analysis 1: Comparison: Febuxostat vs Allopurinol; Test type: Superiority or Other; p = 1.0000, Chi-squared; Relative risk = 0.994, 95% CI 2-sided [0.9691 to 1.0199]

6. Other Pre Specified Outcome: Treatment Emergent Signs or Symptoms (TESS)
Description: Incidence, severity, seriousness and treatment-causality of TESS
Time Frame: 14 ± 2 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 ± 2 days
Description: Analysed for the Safety Population (all patients who received the study drug)
Arm/Group | Febuxostat | Allopurinol
Serious Adverse Events (participants affected / at risk) | 21/173 | 6/173
Other Adverse Events (participants affected / at risk) | 116/173 | 112/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat (N=173) | Allopurinol (N=173)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat (N=173) | Allopurinol (N=173)
Anaemia (Blood and lymphatic system disorders) | 38 (48) | 25 (31)
Leukopenia (Blood and lymphatic system disorders) | 25 (26) | 27 (27)
Neutropenia (Blood and lymphatic system disorders) | 30 (32) | 40 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (28) | 19 (20)
Constipation (Gastrointestinal disorders) | 14 (16) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 16 (21) | 11 (13)
Nausea (Gastrointestinal disorders) | 22 (25) | 21 (23)
Vomiting (Gastrointestinal disorders) | 10 (11) | 12 (12)
Mucosal inflammation (General disorders) | 11 (11) | 3 (3)
Pyrexia (General disorders) | 23 (25) | 18 (21)
Platelet count decreased (Investigations) | 9 (9) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (7) | 9 (10)
Hyperphosphataemia (Metabolism and nutrition disorders) | 9 (9) | 4 (4)
Headache (Nervous system disorders) | 13 (14) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less